CLINICAL TRIAL: NCT04454970
Title: Safe Access for Bladder Entry in Transgender Men Following Penile Reconstruction: a Randomised Controlled Trial
Brief Title: Safe Access for Bladder Entry in Transgender Men Following Penile Reconstruction
Acronym: SAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: St Peter's Andrology Centre (Unknown); University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 124568
Record Dates: First submitted 2019-07-16; First posted 2020-07-02 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Transgenderism; Catheter Related Complication
Keywords: urethral catheterisation; phalloplasty; penile reconstruction; transgender
MeSH Terms: conditions — Transsexualism

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant
Masking Description: Participants are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Urethral catheterisation device (UCD) (Experimental): First attempt of urethral catheterisation using the Urethrotech(R) Urethral catheterisation device (UCD)
  Interventions: Device: Urethrotech Urethral catheterisation device (UCD)
- Bardia Aquafil Foley catheter (Active Comparator): First attempt of urethral catheterisation using the Bardia Aquafil Foley catheter
  Interventions: Device: Bardia Aquafil long term catheter

INTERVENTIONS:
Device: Urethrotech Urethral catheterisation device (UCD) — Urethral indwelling catheter
  Other Names: UCD-0035-090-0016
  Arms: Urethral catheterisation device (UCD)
Device: Bardia Aquafil long term catheter — Urethral indwelling catheter
  Other Names: 165814UK
  Arms: Bardia Aquafil Foley catheter

SUMMARY:
Inserting a urinary catheter in transgender men following penile reconstruction is difficult and usually requires specialist input. Specialist input may not always be readily available and clinicians may resort to suprapubic catheterisation with the associated risk of injury to the bowel or blood vessels. There is a need for an evidence-based protocol to guide clinicians faced with having to catheterise one of these patients. The investigators will evaluate how successful a specialised catheter (Urethrotech UCD®) is compared with a standard Foley catheter for catheterisation of these patients. The Urethrotech UCD® is already used for difficult catheterisation in cisgender men. Transgender men undergoing insertion of an inflatable penile prosthesis under general anaesthesia will be recruited and randomly assigned to have either the Urethrotech UCD® or Foley catheter for the first attempt at urethral catheterisation (required for standard care). If unsuccessful, flexible cystoscopy will be performed and a Foley catheter will be inserted over a guidewire. The catheter is generally removed the next day prior to discharge from hospital. Patients will be followed-up in 30 days by phone.

DETAILED DESCRIPTION:
The only patients eligible are transgender men following penile reconstruction undergoing insertion of an inflatable penile prosthesis under general anaesthesia. Patients will be identified by the theatre booking lists at St Peter's Andrology and will be contacted by phone. The trial will be discussed and any concerns addressed. The patient information sheet will be emailed to them (or posted by mail, if preferred by the patient). Patients will be given at least 24 hours to consent to participate in the trial. As much time as possible will be given to consider the information provided.

The study sites (University College London Hospital, The London Clinic and King Edward VII's Hospital) are where the operations for insertion of inflatable penile prosthesis are performed. The sites will not play any other role in the study and equipment for the study will be brought to the hospitals as required.

The consent form will be signed on the morning of the procedure by the patient. Patients who consent to participate in the study will be randomly assigned to having either a Urethrotech UCD or a Bardia Aquafil Foley catheter for their first attempt at urethral catheterisation. If unsuccessful, a flexible cystoscopy (telescopic examination) will be performed and a guidewire passed directly into the bladder. A Foley catheter will then be passed over the wire, into the bladder.

Following surgery, patients will be admitted overnight and the catheter removed the next day followed by discharged. After 30 days, patients will be followed-up by phone.

All data will be kept in a password protected document and no data or intellectual property will be transferred to other research groups although there may be future need to share deidentified data with other groups. All study activities will be performed by the research group.

ELIGIBILITY:
Inclusion Criteria:

* Female to male transgender men following penile reconstruction
* On waiting list for insertion of inflatable penile prosthesis
* Willing and able to provide written informed consent

Exclusion Criteria:

* Transgender men prior to undergoing penile reconstruction
* Cisgender men or women
* Known urethral fistula or stricture that has not been treated
* Declines to be enrolled in trial
* Does not require a urethral catheter for clinical reasons
* Urinary tract infection

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender
Enrollment: 19 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-03-04 (Actual)

PRIMARY OUTCOMES:
Rate of successful catheterisation of the bladder | 15 minutes
  Rate of successful catheterisation is defined by the appearance of urine from the catheter following insertion

SECONDARY OUTCOMES:
Number of passes required prior to successfully catheterising the bladder | 15 minutes
  Number of passes of the integrated guidewire of the urethral catheterisation device or the Bardia Aquafil catheter required in order to catheterise the bladder
Rate of successful catheterisation using flexible cystoscopy into the bladder | 30 minutes
  Rate of successful catheterisation is defined by the appearance of urine from the catheter following insertion
Complication rate | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: David J Ralph, MBBS, MS, Principal Investigator — University College London Hospitals Foundation NHS Trust
Locations (1):
- New Victoria Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bugeja S, Mistry K, Yim IHW, Tamimi A, Roberts N, Mundy AR. A new urethral catheterisation device (UCD) to manage difficult urethral catheterisation. World J Urol. 2019 Apr;37(4):595-600. doi: 10.1007/s00345-018-2499-9. Epub 2018 Sep 24. PMID 30251050
- [Result] Saint S, Trautner BW, Fowler KE, Colozzi J, Ratz D, Lescinskas E, Hollingsworth JM, Krein SL. A Multicenter Study of Patient-Reported Infectious and Noninfectious Complications Associated With Indwelling Urethral Catheters. JAMA Intern Med. 2018 Aug 1;178(8):1078-1085. doi: 10.1001/jamainternmed.2018.2417. PMID 29971436